CLINICAL TRIAL: NCT01768390
Title: Caries-preventive Effectiveness of a Dentifrice Containing 5.000 Ppm Fluoride - a Randomized Controlled Trial in Adolescents With Fixed Orthodontic Appliances
Brief Title: Caries-preventive Effect of a Dentifrice Containing 5,000 Ppm Fluoride in Orthodontic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Svante Twetman, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 417/2007; 1212 (Other: Copenhagen University)
Record Dates: First submitted 2013-01-04; First posted 2013-01-15 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Dental Caries
Keywords: caries; prevention; orthodontics; fixed appliances; adolescents
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5000 Test (Experimental): Twice daily use of a toothpaste containing 5,000 ppm fluoride
  Interventions: Other: toothpaste containing 5,000 ppm fluoride
- 1450 GCP (Active Comparator): Twice daily use of a toothpaste containing 1,450 ppm fluoride
  Interventions: Other: 1450 GCP

INTERVENTIONS:
Other: toothpaste containing 5,000 ppm fluoride — 1 cm tootpaste twice daily during 2 minutes
  Arms: 5000 Test
Other: 1450 GCP — Twice gaily toothbrushing with normal adult toothpaste containing 1450 ppm F representing good clinical practice
  Arms: 1450 GCP

SUMMARY:
AIM: To evaluate the efficacy of daily tooth brushing with high concentrated fluoride dentifrice on white spot lesion (WSL) formation in adolescents during treatment with fixed orthodontic appliances (FOA).

The null hypothesis is that neither incidence nor severity of lesions would differ from a control group using standard fluoride dentifrice.

SUBJECTS AND METHODS: 420 healthy consecutive 11-16 year-old patients referred to 4 Orthodontic Specialist Clinics are randomized to use either a dentifrice containing 5.000 ppm fluoride or a regular dentifrice with 1.450 ppm sodium fluoride. To be eligible for inclusion, the patients are scheduled for bimaxillary treatment with FOA for an expected duration of at least 1 year. All are instructed to use 0.25 gram dentifrice and brush their teeth during 2 minutes twice daily during the entire period of treatment. Before bonding, and after polishing with a rubber cup and non-fluoride pumice paste, 3 digital photos of the maxillary incisors, canines and premolars are taken. At debonding, remaining composite material on the surfaces is removed with a slow rotating carbide bur followed by polishing with a rubber cup and pumice paste. A new series of frontal and lateral digital photos is thereafter exposed.

The primary outcome measure is the incidence and severity of WSL as registered separately by two blinded experienced and calibrated clinicians according to a validated index. A random sample of 50 cases is re-assessed to check intra- and inter-examiner reliability. The intervention is indended run throughout the full duration of the orthodontic treatment, varying between 18 and 24 months.

DETAILED DESCRIPTION:
not desired

ELIGIBILITY:
Inclusion Criteria:

* healthy
* bi-maxillary treatment with fixed orthodontic appliances for at least 1 year

Exclusion Criteria:

* poor oral hygiene (not being able to brush their teeth)
* recent high caries activity

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2008-01; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
White spot lesion incidence | up to 24 months (at debonding of ortodontic appliances)
  Clinical scoring according to validated index

SECONDARY OUTCOMES:
white spot lesion severity | up to 24 months (at debonding of orthodontic brackets)
  clinical scoring according to a validated index

CONTACTS AND LOCATIONS:
Overall Officials: Svante HA Twetman, professor, Principal Investigator — University of Copenhagen
Locations (1):
- Halland Hospital, Halmstad, Sweden